CLINICAL TRIAL: NCT03633929
Title: mHealth for Patient Self-Management of Opioid Use Disorder
Status: Completed | Type: Observational
Sponsor: Biomedical Development Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-1-100-OUD
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- KIOS OUD
  Interventions: Other: KIOS OUD

INTERVENTIONS:
Other: KIOS OUD — Study Participants will evaluate software known as KIOS-OUD

SUMMARY:
Twenty individuals diagnosed with opioid use disorder (OUD) will be recruited to participate in a beta test to demonstrate feasibility of using an online tool to help them better self-manage their recovery.

DETAILED DESCRIPTION:
Participants will be enrolled in a 4-week single group pre-post evaluation. All participants will attend a two hour orientation to complete baseline assessments, learn how to access and use the software, and participate in a training session. Study participants will be asked to complete assessments online at least three times per week, but no more than once daily. The software may still be accessed by participants as many times as desired to review advice and graphs. After the four week evaluation phase, participants will return for a two hour debriefing and completion of assessment surveys. This approach permits users to be adequately trained while also evaluating the software within their typical environment rather than in a lab setting.

ELIGIBILITY:
Inclusion Criteria:

1. male or female outpatients 18 years of age or older;
2. opioid use disorder as assessed by MINI 6.0;
3. currently stable in OUD outpatient treatment for 4 weeks or longer; and
4. ability to access KIOS-OUD via computer, smartphone, or tablet.

Exclusion Criteria:

1. are unwilling or unable to comply with study requirements;
2. have a major untreated psychiatric illness (e.g., schizophrenia, bipolar disorder) or suicidality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty individuals diagnosed with opioid use disorder
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karla Ramirez, LCSW, Principal Investigator — Consultant
Locations (2):
- United States (2):
  - Biomedical Development Corporation, San Antonio, Texas
  - Community Medical Services, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will share data according to NIMH expectations
Supporting Information: Analytic Code
Time Frame: within 6 months of study completing
URL: https://grants.nih.gov/grants/guide/notice-files/not-mh-14-015.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from private opioid recovery clinics. Recruitment began July 1, 2020 through August 13, 2020
Pre-assignment Details: Participants attended an online orientation on Zoom to learn how to access and use KIOS and participate in a training session.
Period: Overall Study
Arm/Group | KIOS OUD
Started | 19
Completed | 15
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Did not login to software. Did not participate | 3

BASELINE CHARACTERISTICS:
Groups:
- Beta Test: All study participants used KIOS in a beta test to demonstrate feasibility of the software.
Arm/Group | Beta Test
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Usability Score
Description: The Systems Usability Scale-Modified, a single-factor, 10-item self-report scale was used to evaluate participants' subjective experience using the software. Systems Usability Scale yields a single number representing a composite measure of the overall usability of the system being studied. Systems Usability Scale scores have a range of 0 to 100, with higher scores representing a better outcome. Systems in early development may expect to have a rating of 30, while more mature systems should rate between 60 - 80.
Time Frame: Usability was assessed at end of the study, at 4 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | KIOS OUD
Number analyzed (Participants) | 15
score on a scale | 89.5 (9.2)

2. Secondary Outcome: Opioid Use
Description: The total number of times opioid use was reported through the application pooled across all participants, self-reported in app.
Time Frame: 4 weeks
Measure: Number; unit: reported use of opioids
Arm/Group | KIOS OUD
Number analyzed (Participants) | 15
reported use of opioids | 1

3. Secondary Outcome: Mean Change in Depression Score From Baseline
Description: The Patient Health Questionnaire will be used to measure depression. This instrument is a nine question survey regarding depression in which patients answer on a 4 point scale (Not at all, Several days, More than half the days, or Nearly every day). A 0-3 number is applied to each answer and multiplied by the number of answers (9), and then summed. Scores range from 0-27 with higher scores indicative of greater depression severity.
Time Frame: This instrument was administered at baseline and at the end of the study (4 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | KIOS OUD
Number analyzed (Participants) | 15
scores on a scale | -1.00 (5.06)

4. Secondary Outcome: Change in World Health Organization Quality of Life Assessment From Baseline
Description: The World Health Organization Quality of Life Assessment - Brief version will be used to measure quality of life pre and post study. This instrument is an abbreviated generic Quality of Life Scale developed through the World Health Organization. This is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely". The instrument covers four domains each with specific facets: Physical Health, Psychological, Social Relationships, and Environment. The domain scores are reported individually. The total range for each domain score is from 4 - 20. Higher values represent a better outcome.
Time Frame: This instrument was issued at baseline and at the end of study (4-weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | KIOS OUD
Number analyzed (Participants) | 15
scores on a scale
  Physical Domain | 0.11 (2.45)
  Psychological Domain | 1.29 (2.86)
  Social Domain | 0.36 (3.11)
  Environment Domain | 0.67 (2.87)

5. Secondary Outcome: Mean Change on Patient-entered Data From KIOS App
Description: Patients self-reported in the KIOS app on their craving, depressed mood, anxiety, irritability, absenteeism, conflicts with others, difficulty completing usual activities, difficulty sleeping, restlessness/agitation, and pain. All assessments were made in app on 0-6 visual analog scale with higher scores representing a worse outcome. Results are reported as mean change from baseline to the averages of individual assessment values taken during the final week of the study.
Time Frame: baseline 4-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KIOS OUD
Number analyzed (Participants) | 15
score on a scale
  Craving | -1.01 (1.55)
  Depressed Mood | -1.20 (1.76)
  Anxiety | -1.48 (1.63)
  Absenteeism | -1.05 (1.72)
  Difficulty with usual activities | -1.08 (1.25)
  Conflicts with Others | -1.30 (1.83)
  Irritability | -1.57 (1.69)
  Difficulty Sleeping | -1.33 (1.91)
  Restlessness/Agitation | -1.47 (1.72)
  Pain | -0.47 (1.60)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | KIOS OUD
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03633929/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03633929/SAP_001.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03633929/ICF_002.pdf